CLINICAL TRIAL: NCT03910504
Title: Anaesthesia With or Without Neuromuscular Blocking Agents in Intubation and Intraoperative Nerve-monitoring During Thyroid Surgery: a Feasibility and Safety Pilot Study.
Brief Title: Anaesthesia With or Without Rocuronium in Intubation and Intraoperative Nerve-monitoring During Thyroid Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico Longhini (Other)
Responsible Party: Sponsor-Investigator, Federico Longhini, Associate Professor, University Magna Graecia
Organization: University Magna Graecia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IONM
Record Dates: First submitted 2019-02-18; First posted 2019-04-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Thyroid; Neuromuscular Blockade; Anesthesia Complication; Anesthesia Intubation Complication
MeSH Terms: conditions — Thyroid Diseases | interventions — Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rocuronium 0,3 mg/kg (Active Comparator): One hour before the operation the patient will receive the midazolam from 1 to 5 mg intravenous. After the adequate preoxigenation and denitrogenation, the induction phase will be performed with the propofol 2 mg/kg intravenous bolus (for the sedation). At the same time continues infusion of remifentanyl (up to 1 mcg/kg/min) will guarantee the adequate anaesthesia.
  Patients, who have been randomized to this group, will be obtained single reduced dose of rocuronium (0,3 mg/kg) once intravenous bolus. The dose of rocuronium will be prepared by an external investigator, to leave the anesthesiologist blinded of the group treatment. The drug will be diluited in a syringe with 20 ml of solution.
  Interventions: Drug: Rocuronium 0.3 mg*kg
- No rocuronium (Experimental): One hour before the operation the patient will receive the midazolam from 1 to 5 mg intravenous. After the adequate preoxigenation and denitrogenation, the induction phase will be performed with the propofol 2 mg/kg intravenous bolus (for the sedation). At the same time continues infusion of remifentanyl (up to 1 mcg/kg/min) will guarantee the adequate anaesthesia.
  Patients, who have been randomized to this group, will not receive rocuronium, but normal saline will be administered by the anesthesiologist in charge of the patients. The dose of normal saline (20 ml in one syringe) will be prepared by an external investigator, to leave the anesthesiologist blinded of the group treatment.
  Interventions: Drug: No Rocuronium

INTERVENTIONS:
Drug: Rocuronium 0.3 mg*kg — Patients randomized to the control group will receive rocuronium at 0.3 mg*kg ev bolus at the induction of anesthesia.
  Other Names: Neuromuscular blockade
  Arms: Rocuronium 0,3 mg/kg
Drug: No Rocuronium — Patients randomized to the interventional group will not receive neuromuscular blockade at the induction of anesthesia.
  Other Names: No neuromuscular blockade
  Arms: No rocuronium

SUMMARY:
In this randomized controlled trial the investigators want to assess if, compared to controls, the administration of one single low-dose of rocuronium would increase the occurrence of absent or weak (i.e. amplitude <100 μV) signal at V1 and R1, indicating a residual NMBA activity. In addition, we also recorded: 1) the occurrence of difficult laryngoscopy; 2) the time-to-intubation; 3) the occurrence of difficult intubation; 4) the number of intubation attempts; 5) the intubation failure rate; 6) the need for oxygenation between intubation attempts; 7) the lowest peripheral saturation in oxygen (SpO2); 8) the number of severe desaturations; 9) the time-to-V1 and 10) the number of post-surgical complications.

DETAILED DESCRIPTION:
The lesion of laryngeal nerves is one of the most severe complications, which could be observed during the thyroid and parathyroid surgery. The recent clinical review, relative the problem and based on 27 articles and 25000 patients involved, shows that the incidence of the temporary paralysis of the recurrent laryngeal nerve (RLN) was 9,8%, and the permanent paralysis of the nerve was 2,3%. In the most cases the typical reasons of lesions of RLN are: section, clamping, electrothermic damage, stretching or entrapment of the nerve. The lesions of the RLN could lead to voice disturbance, breathing and swallow alterations. It is also one of the most frequent reasons for legal medicine disputes.

The intraoperative nerve-monitoring (IONM) of the RLN and of the external branch of superior laryngeal nerve (EBSLN) has been suggested as an instrument to limit the risk of post-operative damaging. It was introduced in the 60's, and the method was accepted by surgical community with the great enthusiasm. This technique is based on employment of special electrode, which transmits electrical signal of low amperage and stimulates directly the RLN, evaluating the muscle response. The stimulation of the EBSLN is commonly identified by contractions of cricothyroid muscle. On the other hand, the stimulation of the RLN leads to the response of the relative vocal cord, which could be palpated or observed by means of electromyography (EMG).

For implementation of the good IONM the collaboration between the surgeons and the anaesthesiologists is strongly required, e.g. the vocal cords are been monitored during the operation by means of laryngoscopy or a special endotracheal tube.

The particular role for the anaesthesiologists during the operation is the way of using of muscle relaxants. In fact, long-action agents should be generally avoided to prevent the absence of adequate muscle response, during the IONM.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery of the thyroid with the use of Intra-Operative Neuromuscular Monitoring (IONM)

Exclusion Criteria:

* Patients who suffer from paralysis of vocal cords or diseases of neuromuscular system.
* Patients with a history of allergy to anaesthetic drugs.
* Patients who has a high possibility of difficult intubation due to one the following criteria: a) interdental distance < 20 mm; b) marked upper teeth protrusion (mandibular prognathism), which is not possible to correct; c) thyromental distance ≤ 60 mm; d) Mallampati class 4; e) macroglossia with marked micrognathia; f) fixed neck flection; g) severe scar tissue or post radiation fibrosis of the tongue.
* Patients who has a high possibility of difficult intubation due to two of the following criteria, associated with each other: a) interdental distance < 35 mm; b) moderate prognathism or retrgnathia; c) mentohyoid distance < 40 mm; d) thyromental distance ≤ 65 mm; e) Mallampati class 2-3; f) reduced head-neck flexion and extension; g) Body Mass Index (BMI) > 30 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of absent or weak signal at V1 and R1 (i.e. amplitude <100 μV) | Immediately after vagus and recurrent laryngeal nerve identification
  Record of the vagus (V1) and recurrent laryngeal nerve (R1) with the intraoperative neuromuscular monitoring before the dissection of the thyroid

SECONDARY OUTCOMES:
Time of intubation | Immediately after successful endotrachel intubation
  The time of intubation is intended as the duration from the moment when the anaesthesiologist takes the laryngoscope till the first end-tidal carbon dioxide record
Rate of difficult intubation | Immediately after successful endotrachel intubation
  Difficult orotracheal intubation is defined as an intubation, which requires more than 2 laryngoscopies, which continues more than 10 minutes, or whether it claims the use of alternative devices
Cormack Lehane scale value | Immediately after successful endotrachel intubation
  Evaluation of laryngeal exposition according to Cormack-Lehane (1: Full view of glottis; 2a: Partial view of glottis; 2b: Only posterior extremity of glottis seen or only arytenoid cartilages; 3: Only epiglottis seen, none of glottis seen; 4: Neither glottis nor epiglottis seen)
V1 time | Immediately after vagus identification
  The time passed from the cutaneous incision until the measurement of V1 (pre-dissection stimulation of vagus nerve)
incidence of post-operative complication | At 48 hours from surgery
  The incidence of post-operative complication (paralysis of RLN, hyporparathyroidism, bleeding or infections of surgical site, dysphagia, post-operative lung complications).
Post-dissection vagus stimulation value | Immediately after the complete removal of the thyroid
  Record of the vagus stimulation (V2) with the intraoperative neuromuscular monitoring after the dissection of the thyroid
Post-dissection recurrent nerve stimulation value | Immediately after the complete removal of the thyroid
  Record of the recurrent nerve stimulation (R2) with the intraoperative neuromuscular monitoring at the end of the dissection of the thyroid
Pain assessment | Immediately after the end of the surgery
  Evaluation of postoperative pain by means of the numeric pain rating scale from 0 (no pain) to 10 (maximal severe pain)
Predissection recurrent nerve stimulation value | Immediately after recurrent nerve identification
  Record of the recurrent nerve stimulation (R1) with the intraoperative neuromuscular monitoring before the dissection of the thyroid
Predissection vagus stimulation value | Immediately after vagus identification
  Record of the vagus stimulation (V1) with the intraoperative neuromuscular monitoring before the dissection of the thyroid

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Dipartimento di Scienze Mediche e Chirurgiche, Università Magna Graecia
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, datasets used and analysed during the current study will be available on reasonable request at the corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication
Access Criteria: On reasonable request at the corresponding author